CLINICAL TRIAL: NCT05531188
Title: Efficacy Evaluation and Cutaneous Acceptability of the LIPIKAR Med Product on Subjects With Atopic Dermatitis Study Conduct Under Cosmetic Form
Brief Title: Efficacy Evaluation and Cutaneous Acceptability of the Lipikar Med Product on Subjects With Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: LRP 20003 LIPIKAR
Record Dates: First submitted 2022-07-26; First posted 2022-09-07 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin microbial flora
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we will test the tolerance of a topical product and its efficacy in reducing the atopy crisis duration and severity. The product will be tested alone, in children and adults with acute mild to moderate AD i.e as an alternative to alternative treatments, over 6 weeks.

DETAILED DESCRIPTION:
Atopic dermatitis is a frequent chronic inflammatory skin disease affecting up to 20% of children and 8% of adults in developed countries. The disease is often localized with predilection for the face and limb folds but can be more widespread. AD is a chronic condition with many patterns of natural history the most frequent of which starting during infancy with spontaneous resolution after several years of an evolution characterized by alternance of flares and remissions. Other natural history profiles are also frequent and the disease is prevalent in adults as well, whether as a continuation of pediatric forms or as later onset diseases. Flares and remissions may as well altern in many different ways. AD is often associated with other atopic conditions including asthma, conjunctivitis and rhinitis5. Per se, the disease generates erythematous vesiculous plaques often associated with pruritis1. With time, lesion may become thicker (i.e. lichenified) and pruritus significantly impacts quality of life and sleep quality. The chronic and recurrent evolution is also felt as a burden by many patients and parents.

Taking into account the various signs and symptoms (including itch and sleep disturbance), scores have been developed to properly assess severity and guide treatment, SCORAD being one of them used both in clinical practice and clinical research. Between flares, AD management aims at preventing recurrence by avoiding triggering factors and restoring skin barrier through daily application of emollients. During flares, topical steroids are more often used than calcineurin inhibitors mostly dedicated to sensitive areas (face, folds). More severe or resistant cases deserve phototherapy or systemic immunomodulatory treatments with many new drug candidates under clinical development. Back to topical treatments, many failures are due to improper usage of topical steroids because of corticophobia. As for calcineurin inhibitors, irritation is the main limiting factor10,11. This is where important room remains for new topical treatments with good safety and tolerance profiles leading to proper usage and good observance over time and avoiding as much as possible steroid application. Crisaborole has recently been authorized in the US and JAK inhibitors are currently under investigation which illustrates the actual need. AD pathophysiology is complex and its apprehension evolves over time. Current vision associates genetic background and environmental triggering factors. Three mains factors interact to generate AD namely 1) skin barrier defect, 2) skin inflammation driven by T lymphocytes and 3) dysbiosis through the decrease of skin microbiome diversity and staphylococcus proliferation. All three are deeply interlinked. Focusing on the latter, evidence is available that microbiome is disturbed during AD. Whether this dysbiosis is a cause or a consequence remains sometimes debated, but growing evidence suggests a causative relationship especially through S. aureus proliferation, at least as an aggravative factor. Indeed S. aureus is way more frequent on AD skin with good correlation with AD severity. Some of S aureus virulence factors (superantigens, enterotoxins, alphatoxins, proteases activators production) provide a good rational for it from a mechanistic standpoint. The decrease of the microbiome diversity, the role of which is to avoid pathogens proliferation, may play a role in S. aureus proliferation on AD skin, together with skin barrier and immune defect.

Therefore, making available well tolerated and easy to use topical products avoiding S. aureus proliferation and dysbiosis fully makes sense whether as standalone or companion products both in flares management and prevention of recurrences.

In this study, the sponsor will test a well tolerated topical product including a phage derived recombinant endolysine (Staphefekt®) with a capacity to specifically destroy S aureus regardless of its methicillin sensitivity. The product will be tested alone, in children and adults with acute mild to moderate AD i.e as an alternative to alternative treatments, over 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

Sex: female and male; Age: children from 2 to 17 years old, adults from 18 to 75 years old; Phototype: all phototypes Subjects with atopic dermatitis lesions that does not exceed 400 cm2, the studied area must be of evaluable size; 50% of the subjects having atopic dermatitis lesion mainly on the face and neck; 50% of the subjects having atopic dermatitis lesion mainly on the body (folds, trunk limbs, etc.); Subject with mild to moderate atopic dermatitis, IGA 2 (75% of the subjects) to 3 (25% of the subjects); Locally on the lesional area (face/ neck or fold): IGA 2 to 3. Subject having given his/her free informed, written consent; Subject willing to adhere to the protocol and study procedures.

Exclusion Criteria:

Subjects presenting symptoms of COVID - 19 (moderate fever, dry cough, and other symptoms as described by the World Health Organisation); Subjects with a temperature higher than 37.5°C; Subject having been tested positive for COVID-19 and without a medical certificate from the Government; For women: pregnant or nursing woman or woman planning to get pregnant during the study; Children less than two years old; Severe atopic dermatitis (IGA>3); Presenting lichenification 1 or 2 for the 25% of subjects with IGA 3; Presenting with another dermatological condition that could interfere with clinical evaluation; Presenting with a previous history of allergy to cosmetic products; Current and past (last 2 weeks) systematic use of topical or systemic antihistamines, topical or systemic steroids, cyclosporin A and other immunosuppressant, naltrexone, paroxetin, fluvoxamine, amitriptylin;

Wash-out treatment for prior or concomitant therapy:

Subjects using systemic anti-inflammatory or immunomodulatory treatments, UV phototherapy or topical high-potency corticosteroids one month prior to study inclusion; Subjects using topical medium-potency corticosteroids, topical calcineurin inhibitors, topical retinoids, topical antimycotic treatments, oral antibiotics for infected AD, within 2 weeks prior to study inclusion; Subjects having used topical low-potency corticosteroids or topical antibacterial medications within 1 week prior to Day 1; Use of topical or systemic treatment during the previous weeks liable to interfere with the assessment of the cutaneous acceptability/efficacy of the study product; Subject having undergone a surgery under general anesthesia within the previous month; Excessive exposure to sunlight or UV-rays within the previous month; Current infection of AD lesions requiring antimicrobial therapy; Current acute or chronic condition unless considered clinically irrelevant and stable by the investigator ; Inability to provide informed consent or comply with study instructions; Subject enrolled in another clinical trial during the study period.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study took place in Mauritius. Population comes from a database of subjects registered as suffering from DA. Further to facilitate recruitment, agents were appointed to look out for subjects presenting the required condition
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Evolution in Investigator Global Assessment (IGA) | Day 0, Day 7, Day 14, Day 21 and Day 42
  The dermatologist uses the IGA score to evaluate the overall appearance of the lesions and evaluation of time of resolution of the studied lesion. A decrease is expected in the number and percentage of subjects who evolve from Clear to almost Clear (IGA 0-1) at each visit
Evolution in score of atopic dermatitis | Day 0, Day 7, Day 14, Day 21 and Day 42
  The dermatologist uses the global local SCORAD score to evaluate the overall appearance of all the lesions. The following signs are recorded on all the application zones:erythema, oedema/papulation, oozing/crusting, excoriation, lichenification, xerosis.
  For each sign on the application zone:
  - intensity will be reported using the following 4-point scale and their respective mean scores will be noted.
  A decrease in the global score is the expected result. The parameter results will be evaluated individually and must decrease

SECONDARY OUTCOMES:
Evolution in Patient Oriented SCORAD (PO-SCORAD) | Day 0, Day 7, Day 14, Day 21, Day 28 and Day 42
  Subject/Parent assess the PO SCORAD themselves using the PO SCORAD scale. Assessment will be performed by analyzing the evolution of the PO SCORAD from baseline. A decrease in the PO SCORAD is the expected result.
Evolution in Surface area affected | Day 0, Day 7, Day 21 and Day 42
  Centimetric measurements (length and breadth) of the studied lesion are done with a measuring tape. Repositioning masks will be done to identify the studied area on next kinetics. The results will be analyzed for a decrease in the surface area of the studied lesion.
Evolution in Clinical scoring of pain | Day 0, Day 7, Day 14, Day 21, Day 28 and Day 42
  The autoscoring of pain is performed by subjects themselves on a Visual Analogic Scale (VAS) of 10 cm
Evolution in Evolution in Patient Oriented Eczema Measure (POEM) | Day 0, Day 7, Day 14, Day 21 and Day 42
  The POEM is a validated, reliable and simple tool for measuring atopic eczema severity in adults and children. The subjects/parents fill in a POEM questionnaire
Evolution in Quality of life questionnaire (DLQI &CDLQI) | Day 0, Day 7, Day 21 and Day 42
  The subjects or subjects parents answer to a DLQI (Dermatology Life Quality Index) or CDLQI (Children Dermatology Life Quality Index) questionnaire consisting of 10 questions concerning their perception of the impact of atopic dermatitis on different aspects of their health-related quality of life over the last week. Improvement is characterized by a decrease in the score.
Evolution in global cutaneous acceptability by the subject/parent | Day 7, Day 14, Day 21, Day 28 and Day 42
  The subject/parent assesses the global cutaneous acceptability of the investigational product using the 5-point scale.
  0: bad
  1. light
  2. moderate
  3. good
  4. very good.
  Descriptive statistics will be done where the frequency and percentage frequency will be calculated. The percentage of subjects with aggravation, no change and improvement will be calculated.
Evolution in global cutaneous acceptability by the dermatologist | Day 7, Day 14, Day 21, Day 28 and Day 42
  The dermatologist investigator assesses the global cutaneous acceptability of the investigational product using the 5-point scale.
  0: bad
  1. light
  2. moderate
  3. good
  4. very good.
  Descriptive statistics will be done where the frequency and percentage frequency will be calculated. The percentage of subjects with aggravation, no change and improvement will be calculated.
Evolution in global efficacy by the subject/parent | Day 7, Day 14, Day 21, Day 28 and Day 42
  The subject/parent assesses the global cutaneous acceptability and efficacy of the investigational product using the 4-point scale.
  0: not effective
  1. little effective
  2. effective
  3. very effective.
  Descriptive statistics will be done where the frequency and percentage frequency will be calculated. The percentage of subjects with aggravation, no change and improvement will be calculated.
Evolution in global efficacy by the dermatologist | Day 7, Day 14, Day 21, Day 28 and Day 42
  The dermatologist investigator assesses the global cutaneous acceptability and efficacy of the investigational product using the 4-point scale.
  0: not effective
  1. little effective
  2. effective
  3. very effective.
  Descriptive statistics will be done where the frequency and percentage frequency will be calculated. The percentage of subjects with aggravation, no change and improvement will be calculated.
Illustrative photographs | Day 0, Day 7, Day 14, Day 21 and Day 42
  The digital camera used is a camera of the type Nikon D7100. Standardized photo acquisition with use of a tripod to facilitate repositioning at all visits will be performed to get illustrative photographs. The photographs are taken in standardized, indirect light. Aperture, speed and distance of the camera are also standardized
Photographs using COLORFACE® | Day 0, Day 7, Day 14, Day 21 and Day 42
  The ColorFace© acquisition system is a dedicated solution for standardized imaging in the clinical study setting for evaluation of a clinical effect or for a screening phase.
  This innovative solution is based on a high-resolution sensor to obtain images of an exceptional quality.
Swabbing | Day 0, Day 42
  Skin microbial flora swabbing are done on one affected zone and on one none affected zone, according to the swabbing protocol
Subjective evaluation questionnaire | Day 21, Day 42
  A subjective evaluation questionnaire is filled in by the subjects to subjectively evaluate the properties of the studied product, its global efficacy and its future use

CONTACTS AND LOCATIONS:
Overall Officials: Aslham Doarika, Principal Investigator
Locations (1):
- Insight Research, Quatre Bornes, Mauritius